CLINICAL TRIAL: NCT01505803
Title: The Effect of a Nutritional Supplement on Cardiometabolic, Inflammatory, and Oxidative Stress Markers in Individuals With Type 2 Diabetes Mellitus: a Pilot Study
Brief Title: The Effect of a Nutritional Supplement in Individuals With Type 2 Diabetes Mellitus: a Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HREC 12392
Record Dates: First submitted 2011-10-25; First posted 2012-01-09 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance
Keywords: Type 2 diabetes mellitus; Dietary supplements; Hyperglycemia; Insulin resistance; Dyslipidemia; Inflammation; Oxidative stress; Zinc; Omega 3
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Hyperglycemia; Dyslipidemias; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Zinc supplement (Active Comparator)
  Interventions: Dietary Supplement: Zinc supplements; Dietary Supplement: Placebo supplements
- Omega 3 supplement (Active Comparator)
  Interventions: Dietary Supplement: Omega 3 supplements; Dietary Supplement: Placebo supplements
- Zinc and omega 3 supplements (Active Comparator)
  Interventions: Dietary Supplement: Zinc supplements; Dietary Supplement: Omega 3 supplements
- Placebo supplement (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo supplements

INTERVENTIONS:
Dietary Supplement: Zinc supplements — Participants will receive 40 mg of zinc each day for 12 weeks.
  Arms: Zinc and omega 3 supplements; Zinc supplement
Dietary Supplement: Omega 3 supplements — Participants will receive 2 g of omega 3 fatty acids each day for 12 weeks.
  Arms: Omega 3 supplement; Zinc and omega 3 supplements
Dietary Supplement: Placebo supplements — Participants will receive placebo supplements each day for 12 weeks.
  Arms: Omega 3 supplement; Placebo supplement; Zinc supplement

SUMMARY:
Diabetes Mellitus (DM) is a major risk factor for cardiovascular disease, with 50% of diabetes-associated deaths being attributed to cardiovascular complications. The characterising features of DM include: the presence of chronic hyperglycaemia, consequent upon decreased secretion or action of insulin; dyslipidaemia; and enhanced levels of oxidative stress and inflammation. Zinc and omega 3 polyunsaturated fatty acids have been shown to influence each of these outcomes via several mechanisms. This pilot study will examine the effect of nutritional supplements containing zinc and omega 3 on these outcomes in a population with type 2 DM.

DETAILED DESCRIPTION:
The prevalence of type 2 DM and related-complications continues to increase. Diet is a significant factor in the aetiology of type 2 DM. Intakes of zinc and omega 3 fatty acids may modulate glycaemic control, lipid metabolism, and inflammatory processes in the disease. Zinc is involved in many biological processes that include enzyme action, stabilisation of cell membranes, regulation of gene expression, and cell signalling. Zinc supplementation has been demonstrated to improve glycaemic control in both animals and humans. The normalising effect of zinc on glucose homeostasis may relate to its involvement in insulin metabolism. Zinc functions in the synthesis, storage, secretion, and action of insulin. Omega-3 also enhances glycaemic control and dietary supplementation with omega-3 polyunsaturated fatty acids has been shown to improve insulin sensitivity in subjects with DM. Both zinc and omega-3 function to mediate lipid metabolism. Zinc supplementation has been found to be associated with a beneficial increase in HDL cholesterol concentrations in individuals with type 2 DM. The mechanism may again involve insulin, which has been proposed as an independent predictor of plasma HDL. Omega-3 directly activates transcription factors that regulate lipid metabolism and is known to decrease serum triglyceride levels in DM. Zinc appears to beneficially impact oxidative stress-related parameters in DM via a range of mechanisms, including the regulation of copper,zinc superoxide dismutase, metallothionein, NF-κB and nitric oxide signaling. The purpose of this pilot study is to explore the effect of zinc and omega 3 supplementation on hyperglycaemia, dyslipidaemia, chronic inflammation, and oxidative stress in a population with type 2 DM.

This study will recruit 48 postmenopausal women with type 2 DM. Participants will be randomly allocated to one of 4 groups for a period of 12 weeks: placebo, zinc, omega 3, or zinc + omega 3 supplementation. Usual dietary intake will be assessed before and after the trial period using 2-day estimated food records, which will be checked by a research dietitian. Blood samples will be collected from all participants at the start of the intervention (week 0) then at 4 weekly intervals (weeks 4, 8, 12) by qualified phlebotomists. Blood samples will be analysed for plasma zinc, plasma lipids and fatty acids, markers of inflammation and oxidative stress, and indicators of glycaemic control. An aliquot of blood will also be used for the measurement of zinc transporter mRNA levels utilising real-time quantitative PCR techniques.

ELIGIBILITY:
Inclusion Criteria:

* Female, postmenopausal
* Type 2 diabetes (controlled by diet and lifestyle; or oral hypoglycaemic medication (i.e. metformin) for not more than 7 years)
* Normal Glomerular Filtration Rate (GFR) and normal microalbumin/creatine ratio
* No nutritional supplements in the 6 weeks prior to the trial & continuing through the trial period
* Non-smoking

Exclusion Criteria:

* Diagnosed with current major illness (renal disease, significant cardiovascular disease, gastrointestinal disorders, cancer, or other significant disorder likely to interfere with zinc metabolism)
* Taking medications that are likely to interfere with zinc metabolism

Min Age: 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Plasma lipids (total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides) | 12 weeks
Glycaemic control (glucose, insulin, HbA1c) | 12 weeks
Inflammation & oxidative stress (CRP, TNF-α, IL-1, IL-2, IL-6, IL-10 F2 isoprostanes, NF-κB, MPO, other) | 12 weeks

SECONDARY OUTCOMES:
Zinc transporter mRNA expression in peripheral blood mononuclear cells | 12 weeks
Plasma zinc | 12 weeks
Plasma fatty acids | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Samir Samman, Principal Investigator — University of Sydney; Meika Foster, Principal Investigator — University of Sydney
Locations (1):
- University of Sydney, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Foster M, Petocz P, Samman S. Effects of zinc on plasma lipoprotein cholesterol concentrations in humans: a meta-analysis of randomised controlled trials. Atherosclerosis. 2010 Jun;210(2):344-52. doi: 10.1016/j.atherosclerosis.2009.11.038. Epub 2009 Nov 29. PMID 20034629
- [Background] Foster M, Samman S. Zinc and redox signaling: perturbations associated with cardiovascular disease and diabetes mellitus. Antioxid Redox Signal. 2010 Nov 15;13(10):1549-73. doi: 10.1089/ars.2010.3111. PMID 20568953
- [Background] Foster M, Hancock D, Petocz P, Samman S. Zinc transporter genes are coordinately expressed in men and women independently of dietary or plasma zinc. J Nutr. 2011 Jun;141(6):1195-201. doi: 10.3945/jn.111.140053. Epub 2011 Apr 13. PMID 21490290